CLINICAL TRIAL: NCT03656055
Title: Study of the Link Between Retinal Atrophy and Demyelinating Inflammatory Processes on Visual Pathways in Relapsing Multiple Sclerosis in Magnetic Resonance Imaging and Optical Coherence Tomography
Brief Title: Analysis of Neurodegenerative Process Within Visual Ways In Multiple Sclerosis
Acronym: VWIMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_32; 2017-A00194-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-08-27; First posted 2018-09-04 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: MRI; axonal loss; MS; OCT
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will interest in the pathophysiology of silent retinal axonal loss in multiple sclerosis. Recent studies have suggested that silent retinal axonal loss (no past history of optic neuritis [ON]) may be due to inflammatory lesions within the optic radiations and a transsynaptic degenerative process. The objective is to measure the exact role of silent optic nerve lesion in the occurrence of silent retinal axonal loss by performing OCT, brain and optic nerve MRI in a cohort of patients without recent disease activity.

DETAILED DESCRIPTION:
This study will interest in the neurodegenerative process reported in multiple sclerosis within the visual ways.

Symptomatic and asymptomatic retinal axonal loss in multiple sclerosis (MS) have largely been described. Many recent optical coherence tomography (OCT) studies have suggested that subclinical retinal axonal loss (no past history of optic neuritis [ON]) observed in MS mainly due to inflammatory and demyelinating lesions within the optic radiations and a retrograde transsynaptic degenerative process. None of these studies clearly tried to investigate the role of asymptomatic optic nerve lesion(s) in subclinical retinal axonal loss occurence.

The main objective of the study is to measure the exact role of silent optic nerve lesion in the occurrence of silent retinal axonal loss by performing OCT, brain and optic nerve MRI. The study will focus on a cohort of patients without recent disease activity in order to exclude or minimize the risk of recent and old lesion occurence on the visual ways, which could be a bias in our analysis.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Remitting Multiple Sclerosis (RRMS) patients treated by natalizumab for more than 6 months
* JohnCunninghamVirus (JCV) index < 0.9
* patients followed in our MS center from the beginning of the disease

Exclusion Criteria:

* ophthalmologic diseases
* diabetes mellitus
* contra-indication to MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RRMS treated by natalizumab for more than 6 months in order to measure patients with a lower risk of relapse
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Study of asymptomatic retinal atrophy in multiple sclerosis and asymptomatic optic nerve demyelinating lesion | Day 1 (cross-sectional study)
  The temporal peripapillary Retinal Nerve Fiber Layer thickness (pRNFL; quantitative data) measured on optical coherence tomography will evaluate asymptomatic retinal atrophy
  Presence of subclinical optic nerve lesion will be assessed on optic nerve MRI (3D-double inversion recovery sequence; Y/N; qualitative data) and according to clinical information (past history of optic neuritis [ON] or not). It will enable investigators to define 3 eyes' groups: eyes' group with symptomatic optic nerve lesion (ON eyes), eyes' group with asymptomatic optic nerve lesion (NON eyes with asymptomatic lesion) and eyes' group without symptomatic or asymptomatic lesion (NON eyes without lesion).
  Investigators will proceed to comparison of temporal pRNFL between NON eyes with asymptomatic lesion and NON eyes without lesion

SECONDARY OUTCOMES:
Evaluation of the link between asymptomatic retinal atrophy in multiple sclerosis and intensity of demyelinating process all along the optic ways (from the retina to the visual cortex) | Day 1 (cross-sectional study)
  Within NON eyes, investigators will evaluate the imaging parameters on the optic ways which is/are significantly and independently associated to temporal pRNFL (multivariate analysis)
  MRI parameters parameters included will be: length of asymptomatic optic nerve lesion; presence of lesion on chiasma, presence of lesion on optic tracts, T2 lesion burden on optic radiations, fractional anisotropy in optic radiations, volume of primary visual cortex
Evaluation of the link between symptomatic retinal atrophy in multiple sclerosis and intensity of demyelinating process all along the optic ways (from the retina to the visual cortex) | Day 1 (cross-sectional study)
  Within ON eyes, investigators will evaluate the imaging parameters on the optic ways which is/are significantly and independently associated to temporal pRNFL (multivariate analysis)
  MRI parameters parameters included will be: length of subclinical optic nerve lesion; presence of lesion on chiasma, presence of lesion on optic tracts, T2 lesion burden on optic radiations, fractional anisotropy in optic radiations, volume of primary visual cortex
Evaluation of the link between retinal atrophy and visual connectivity | Day 1 (cross-sectional study)
  Within all eyes (ON eyes + NON eyes with asymptomatic optic nerve lesion + NON eyes without asymptomatic lesion), investigators will evaluate the link between the mean temporal pRNFL of both eyes (pRNFL; quantitative data) and the strength of visual connectivity (seed based approach on resting state sequence)
Evaluation of the link between visual disability and MRI parameters measuring intensity of demyelinating process all along the optic ways (from the retina to the visual cortex) | Day 1 (cross-sectional study)
  Within all eyes (ON eyes + NON eyes with asymptomatic optic nerve lesion + NON eyes without asymptomatic lesion), investigators will evaluate the MRI parameters significantly and independently associated to visual disability.
  Visual disability will be measured by low contrast vision acuity (2.5%; unit LogMar)
  MRI parameters will be length of subclinical optic nerve lesion; presence of lesion on chiasma, presence of lesion on optic tracts, T2 lesion burden on optic radiations, fractional anisotropy in optic radiations, volume of primary visual cortex

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Outteryck, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodel J, Outteryck O, Bocher AL, Zephir H, Lambert O, Benadjaoud MA, Chechin D, Pruvo JP, Vermersch P, Leclerc X. Comparison of 3D double inversion recovery and 2D STIR FLAIR MR sequences for the imaging of optic neuritis: pilot study. Eur Radiol. 2014 Dec;24(12):3069-75. doi: 10.1007/s00330-014-3342-3. Epub 2014 Aug 23. PMID 25149294
- [Background] Hadhoum N, Hodel J, Defoort-Dhellemmes S, Duhamel A, Drumez E, Zephir H, Pruvo JP, Leclerc X, Vermersch P, Outteryck O. Length of optic nerve double inversion recovery hypersignal is associated with retinal axonal loss. Mult Scler. 2016 Apr;22(5):649-58. doi: 10.1177/1352458515598021. Epub 2015 Jul 30. PMID 26227005
- [Background] Gabilondo I, Martinez-Lapiscina EH, Martinez-Heras E, Fraga-Pumar E, Llufriu S, Ortiz S, Bullich S, Sepulveda M, Falcon C, Berenguer J, Saiz A, Sanchez-Dalmau B, Villoslada P. Trans-synaptic axonal degeneration in the visual pathway in multiple sclerosis. Ann Neurol. 2014 Jan;75(1):98-107. doi: 10.1002/ana.24030. Epub 2014 Jan 2. PMID 24114885
- [Background] Jindahra P, Petrie A, Plant GT. The time course of retrograde trans-synaptic degeneration following occipital lobe damage in humans. Brain. 2012 Feb;135(Pt 2):534-41. doi: 10.1093/brain/awr324. Epub 2012 Feb 1. PMID 22300877
- [Background] Petzold A, Balcer LJ, Calabresi PA, Costello F, Frohman TC, Frohman EM, Martinez-Lapiscina EH, Green AJ, Kardon R, Outteryck O, Paul F, Schippling S, Vermersch P, Villoslada P, Balk LJ; ERN-EYE IMSVISUAL. Retinal layer segmentation in multiple sclerosis: a systematic review and meta-analysis. Lancet Neurol. 2017 Oct;16(10):797-812. doi: 10.1016/S1474-4422(17)30278-8. Epub 2017 Sep 12. PMID 28920886
- [Background] Martinez-Lapiscina EH, Arnow S, Wilson JA, Saidha S, Preiningerova JL, Oberwahrenbrock T, Brandt AU, Pablo LE, Guerrieri S, Gonzalez I, Outteryck O, Mueller AK, Albrecht P, Chan W, Lukas S, Balk LJ, Fraser C, Frederiksen JL, Resto J, Frohman T, Cordano C, Zubizarreta I, Andorra M, Sanchez-Dalmau B, Saiz A, Bermel R, Klistorner A, Petzold A, Schippling S, Costello F, Aktas O, Vermersch P, Oreja-Guevara C, Comi G, Leocani L, Garcia-Martin E, Paul F, Havrdova E, Frohman E, Balcer LJ, Green AJ, Calabresi PA, Villoslada P; IMSVISUAL consortium. Retinal thickness measured with optical coherence tomography and risk of disability worsening in multiple sclerosis: a cohort study. Lancet Neurol. 2016 May;15(6):574-84. doi: 10.1016/S1474-4422(16)00068-5. Epub 2016 Mar 18. PMID 27011339